CLINICAL TRIAL: NCT05797246
Title: A Phase II Study of Bevacizumab in Adults With Recurrent Respiratory Papillomatosis (RRP)
Brief Title: Bevacizumab in Adults With Recurrent Respiratory Papillomatosis (RRP)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001572; 001572-C
Record Dates: First submitted 2023-04-01; First posted 2023-04-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Respiratory Tract Diseases; Neoplasms; Neoplasms by Histologic Type; Neoplasms, Glandular and Epithelial; Neoplasms, Squamous Cell; Tumor Virus Infections; Infections; Virus Diseases; DNA Virus Infections; Pathologic Processes; Disease Attributes; Recurrence; Papilloma; Respiratory Tract Infections; Papillomavirus Infections
Keywords: Human Papilloma Virus; Dose Escalation; laryngotracheal disease; papillomatous disease
MeSH Terms: conditions — Respiratory Tract Diseases; Neoplasms; Neoplasms by Histologic Type; Neoplasms, Glandular and Epithelial; Neoplasms, Squamous Cell; Tumor Virus Infections; Infections; Virus Diseases; DNA Virus Infections; Pathologic Processes; Disease Attributes; Recurrence; Papilloma; Respiratory Tract Infections; Papillomavirus Infections | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Bevacizumab treatment course
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg IV every three weeks for 3 cycles and then every 6 weeks for a total treatment course of 11 cycles for approximately 1 year total.

SUMMARY:
Background:

Recurrent respiratory papillomatosis (RRP) is a rare disease that causes wart-like growths in the airways. These growths come back when removed; some people may need 2 or more surgeries per year to keep their airways clear. Better treatments are needed.

Objective:

To see if a drug called bevacizumab can reduce the number of surgeries needed in people with RRP.

Eligibility:

People aged 18 and older with recurrent RRP; they must need surgery to remove the growths in their airways.

Design:

Participants will be screened. Their ability to breathe and speak will be evaluated. They will have an endoscopy: a flexible tube with a light and camera will be inserted into their nose and throat. They will have a test of their heart function and imaging scans of their chest.

Participants will have surgery to remove the growths in their airways.

Bevacizumab is given through a small tube placed in a vein in the arm. After the surgery, participants will receive 11 doses of this drug: every 3 weeks for 3 doses, and then every 6 weeks for 8 more doses. They will come to the clinic for each dose; each visit will be about 8 hours.

Tissue samples of the growths will be collected after the second treatment; this will be done under general anesthesia.

Participants may undergo apheresis: Blood will be drawn from a needle in an arm. The blood will pass through a machine that separates out the cells needed for the study. The remaining blood will be returned to the body through a second needle.

Follow-up will continue for 1 year after the last treatment.

DETAILED DESCRIPTION:
Background:

* Recurrent respiratory papillomatosis (RRP) is a rare papillomatous disease of the respiratory tract that is caused by Human Papilloma Virus (HPV) types 6 or 11.
* RRP can progress to cause severe voice disturbance, airway compromise, fatal pulmonary lesions, and rarely invasive cancers.
* There is no approved systemic therapy for RRP. Participants require repeated surgical procedures for disease debridement and control.
* Translational research studies have shown high levels of vascularity in papilloma tissue driven in part by high levels of vascular endothelial growth factor (VEGF)-A mRNA, vascular endothelial growth factor receptors (VEGFR)-1 and VEGFR-2 and elevated serum levels of VEGF-A, particularly in cases of aggressive RRP.
* Papillomas are also infiltrated by immunosuppressive myeloid and regulatory T-cells.
* Systemic inhibition of VEGF signaling may reduce VEGF-driven angiogenesis in papillomas and reduce chemotaxis and expansion of immunosuppressive myeloid cells and regulatory T-cells.
* Bevacizumab is a recombinant humanized monoclonal antibody that binds all active forms of VEGF-A.
* Bevacizumab is FDA approved for the treatment of metastatic colorectal cancer, non-small cell lung cancer, metastatic renal cell carcinoma, recurrent glioblastoma, cervical cancer, epithelial ovarian cancer, fallopian tube cancer and primary peritoneal cancer and was selected for its demonstrated activity in a variety of cancers and for its acceptable safety profile.
* Use of systemic bevacizumab in patients with severe and/or tracheal RRP has not been studied prospectively in controlled clinical studies, but clinical safety and activity has been reported in retrospective single institution case series.
* Bevacizumab resistance can develop in cancer patients due to a variety of tumor escape mechanisms that are unlikely to occur in RRP patients with normal endothelial cells, but bevacizumab re-treatment for recurrent RRP has not been evaluated in controlled clinical studies.

Objective:

-To determine the percentage of participants with an increase in their surgery-free interval during treatment with systemic bevacizumab

Eligibility:

* Histologically confirmed diagnosis of RRP
* A history of 2 or more surgeries in the last 12 months in order to control laryngeal and/or tracheal RRP
* At least one of the following:

  * A Derkay score of 8 or greater
  * Pulmonary RRP with disease measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
  * Tracheal involvement with RRP that has required two or more clinical interventions in the last 12 months
  * Tracheostomy
* Age >=18 years old
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1

Design:

* This is a phase II, single arm clinical trial evaluating systemic bevacizumab.
* Participants will receive bevacizumab (10 mg/kg IV) every three weeks for 3 cycles and then every 6 weeks for a total treatment course of 11 cycles for approximately 1 year total.
* Operative examination under anesthesia (EUA) with biopsies for research and possible papilloma debulking for safety will be performed before dose 1, optional EUA for research biopsies may be performed following dose 2 and at cycles 6 and 11.
* Participants may undergo standard-of-care operative EUA with papilloma cleanout during the 1-year treatment period as clinically indicated at the NIH.
* The mean surgery-free interval during the 1-year treatment period will be compared to the mean surgery-free interval in the 12 months prior to treatment.
* Participants will also be assessed for papilloma recurrence and surgery-free interval at 6, 12, 24 weeks and every 3 months after that until 1 year following completion of treatment.
* A total of 20 evaluable participants will be treated on study.
* During the follow up period, up to 15 participants who develop sufficient papilloma recurrence to require a clinical intervention may be re-treated with 11 additional cycles of bevacizumab (10 mg/kg IV) following the same schedule as the initial treatment.
* Prior to the initiation of re-treatment, an optional operative EUA with biopsies for research and possible papilloma debulking for safety may be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >= 18 years old.
* Histologically confirmed diagnosis of RRP.
* Individuals must require procedure(s) to remove papillomatous disease per standard of care.(not required for re-treatment)
* A history of 2 or more surgeries within 12 months prior to treatment initiation in order to control laryngeal and/or tracheal RRP (not required for re-treatment).
* At least one of the following (not required for re-treatment):

  * A Derkay score of 8 or greater
  * Measurable disease per RECIST 1.1 (participants with pulmonary RRP only)
  * Tracheal involvement with RRP that has required two or more clinical interventions in the last 12 months (two or more clinical interventions)
  * Tracheostomy.
* ECOG performance status of 0-1.
* Individuals must have adequate organ and marrow function as defined below:

  * White blood cells (WBC): >2,000/microL
  * Absolute neutrophil count (ANC): >=1,500/microL
  * Hemoglobin: >9.0 g/dL
  * Platelets: >=100,000/microL
  * Total bilirubin: <=1.5 mg/dL, except in participants with Gilbert s Syndrome who must have a total bilirubin less than 3.0 mg/dL
  * Aspartate aminotransferase (AST) /Alanine aminotransferase (ALT): <=2.5 X institutional upper limit of normal (ULN)
  * Creatinine: within normal institutional limits

OR

Creatinine Clearance (CrCl): >=60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal (calculated using the Cockcroft-Gault formula).

* Prothrombin time (PT) /International normalized ratio (INR) and Partial thromboplastin time (PTT): <=1 X institutional ULN. In participants on anticoagulation, coagulation tests should be within a therapeutic range.
* Urinalysis: Urine dipstick < 2+ proteinuria. In participants with >=2+ proteinuria on dipstick urinalysis should undergo a 24-hour urine collection and must demonstrate <=1g of protein in 24 hours to be eligible

  * Individuals must have received their last systemic therapy for RRP > 4 weeks or 5 half-lives, whichever is longer, prior to treatment initiation, except for systemic bevacizumab which must be > 1 year prior to treatment initiation (not applicable for re-treatment)
  * Individuals able to become pregnant and their partners must agree to use highly effective method of contraception (hormonal, intrauterine device (IUD), surgical sterilization ) for the duration of bevacizumab treatment and up to 6 months after completion of bevacizumab treatment. NOTE: Abstinence, defined as no heterosexual sexual intercourse when this is in line with the preferred and usual lifestyle of the individual is also acceptable.
  * Breastfeeding individuals must be willing to discontinue breastfeeding from study treatment initiation through 6 months after bevacizumab treatment discontinuation.
  * All individuals must have the ability to understand and willingness to sign a written informed consent.
  * All individuals must be willing to undergo mandatory biopsy during the study (not applicable for re-treatment).

EXCLUSION CRITERIA:

* History of significant (i.e., active) cardiovascular disease or thromboembolic event: cerebral vascular accident/stroke (within 6 months prior to treatment initiation), myocardial infarction (within 6 months prior to treatment initiation), unstable angina, congestive heart failure (>= New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication as assessed by EKG.
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to treatment initiation.
* Major surgery within 4 weeks prior to treatment initiation.
* Non-healing wound, active ulcer, or untreated bone fracture.
* History of hemoptysis (>2.5 mL of bright red blood per episode) within 1 month prior to treatment initiation.
* Evidence of bleeding diathesis or significant coagulopathy (with or without current therapeutic anticoagulation).
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to treatment initiation.
* Inadequately controlled hypertension (defined as systolic blood pressure (BP) >150 mmHg and/or diastolic blood pressure > 100 mmHg), an average of 3 BP readings on 2 sessions will be used to measure blood pressure if initial reading indicates inadequately controlled hypertension. NOTE: Anti-hypertensive therapy to achieve blood pressures below these parameters is allowed.
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* Persisting toxicity related to prior therapy of Grade >1 per Common Terminology Criteria for Adverse Events (CTCAE) v 5.0. NOTE: alopecia, sensory neuropathy Grade <=2 are acceptable.
* Known active alcohol or drug abuse.
* History of allergy to study drug components.
* Pregnancy (confirmed with Beta-Human chorionic gonadotropin (Beta-HCG) serum or urine pregnancy test in WOCBP performed at screening).
* Uncontrolled intercurrent illness or situation that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
To determine the percentage of participants with an increase in their surgery-free interval during treatment with systemic bevacizumab. | 1 year
  Determined by measuring the mean duration between successive clinically indicated surgeries in the 12 months during treatment for that participant and determining whether that duration is longer than the mean duration between successive clinically indicated surgeries in the 12 months prior to treatment by one month or more. This fraction of participants who are classified as having a success will be reported along with a 95% confidence interval.

SECONDARY OUTCOMES:
Rate of pulmonary RRP partial response (PR) and complete response (CR) by RECIST 1.1 in participants with pulmonary disease. | 6 weeks after completion of treatment
  The fraction of participants with a pulmonary RRP partial response and a pulmonary RRP complete response will be reported in all treated pulmonary participants, along with 95% confidence intervals for each.
Recurrence free interval after treatment | Weeks 6, 12, 24 and remote assessment (if needed)
  Time to recurrence of papillomatous disease after completion of treatment will be recorded and reported descriptively.
The safety of systemic bevacizumab in participants with aggressive RRP | 42 days after the study agent was last administered
  Evaluation of safety will be done as follows: each participant will be evaluated for safety and toxicity, and the fraction of participants experiencing AEs will be reported by type and grade of AE
The rate of papilloma regrowth by determining the percentage of participants with an increase in their surgery-free interval after treatment with systemic bevacizumab | Weeks 6, 12, 24 after completion of treatment, every 3 months after that with the last evaluation performed at 1 year after completion of study treatment
  The rate of papilloma regrowth will be determined by measuring the mean duration between successive clinically indicated surgeries in the 12 months after treatment for that participant and determining whether that duration is longer than the mean duration between successive clinically indicated surgeries in the 12 months prior to treatment by one month or more. This fraction of participants who are classified as having a success will be reported along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Norberg, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001572-C.html